CLINICAL TRIAL: NCT04961957
Title: Waterproof Casting Versus Standard Casting for Short Leg Walking Casts: a Prospective Randomized Controlled Trial
Brief Title: Waterproof Casting Versus Standard Casting for Short Leg Walking Casts
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Casting material has been changed and can no longer proceed with the study.
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, David Tager, Assistant Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2102248177
Record Dates: First submitted 2021-07-07; First posted 2021-07-14 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Ankle Fractures; Foot Fracture; Ankle Sprains; Foot Sprain; Toe-walking; Tendonitis of Foot; Apophysitis; Juvenile
MeSH Terms: conditions — Ankle Fractures; Ankle Injuries

STUDY DESIGN:
Intervention Model Description: This prospective, randomized controlled trial involves the subject being randomized (similar to flipping a coin) by envelope to receive either waterproof padding or non-waterproof padding in their short leg walking cast. The study will take approximately three to seven weeks for the subject to complete (pending date of cast removal).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Waterproof padding (Active Comparator): Waterproof, short leg walking cast for 3-7 weeks
  Interventions: Device: Waterproof padding
- Non-waterproof padding (Active Comparator): Non-waterproof, short leg walking cast for 3-7 weeks
  Interventions: Device: Non-waterproof padding

INTERVENTIONS:
Device: Waterproof padding — Apply waterproof padding to allow for normal bathing and water activities
  Arms: Waterproof padding
Device: Non-waterproof padding — Apply standard padding that does not allow for normal bathing and water activities
  Arms: Non-waterproof padding

SUMMARY:
The purpose of the study is to determine whether the use of waterproof padding in short leg walking casts will lead to an increase in cast-related complications, as compared to the standard non-waterproof casting in children.

DETAILED DESCRIPTION:
This study aims to prospectively examine a group of pediatric patients that receive either a waterproof or non-waterproof short leg cast. From this, we will be able to determine if there are any significant differences between the two groups. If waterproof short leg casts do not cause increased skin breakdown or lead to increases in cast complications and unintended clinic visits, then we can more confidently apply them to pediatric patients, particularly in the summer months when children are more likely to swim.

On application of a waterproof, short leg walking cast, a questionnaire will be distributed to the patient/family to track how many times the cast gets wet. During the application of the cast, materials will be tracked for cost analysis. The subject will return between 3 and 7 weeks for cast removal. On cast removal, the following questionnaires will be completed: cast condition, skin condition, overall patient/family satisfaction, and PROMIS Pediatric Lower Extremity Function - Mobility. Questionnaires will take approximately 5 - 10 minutes to complete. The parent survey regarding how many times the cast got wet will be returned (if applicable). Waterproof and non-waterproof groups will be compared in the basis of cast condition, PROMIS lower extremity survey outcomes, skin condition, overall patient/family satisfaction, number of unintended cast changes or return clinic visits, as well as cost difference.

Outside of the randomization itself, all standard of care procedures or normal practice activities will occur. Each participant will undergo cast application as recommended per standard of care. Study participation does not involve more than minimal risk since everything outside of the randomization is standard of care.

Waterproof and non-waterproof groups will be compared in the basis of cast condition, PROMIS lower extremity survey outcomes, skin condition, overall patient/family satisfaction, number of unintended cast changes or return clinic visits, as well as cost difference. A Chi-Square test will be used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

• Being placed in a short leg walking cast for one of the diagnoses listed below:

* ankle fracture
* foot fracture
* ankle sprain
* foot sprain
* toe-walking
* tendonitis
* apophysitis

Exclusion Criteria:

* Patients with wounds to the foot or ankle prior to cast placement
* Patients with cognitive dysfunction

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Preference for Same Type of Cast (waterproof short leg walking cast) | Upon Cast Removal (3-7 weeks from cast application)
  Proportion of patients who, after treatment, express a preference for the same type of cast.
Preference for Same Type of Cast (non-waterproof short leg walking cast) | Upon Cast Removal (3-7 weeks from cast application)
  Proportion of patients who, after treatment, express a preference for the same type of cast.

CONTACTS AND LOCATIONS:
Overall Officials: David Tager, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No